CLINICAL TRIAL: NCT05404386
Title: The Effect of Mobile Application on Incontinence Symptoms, Compliance With Kegel Exercises, Health Belief, and Quality of Life of Women With Urinary Incontinence
Brief Title: Effect of Mobile Application on Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Pınar Duru, Assistant Professor Doctor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AliCicekli
Record Dates: First submitted 2022-05-28; First posted 2022-06-03 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Urinary Incontinence,Stress; Urinary Incontinence, Urge; Urinary Incontinence, Mixed; Symptoms; Kegel Exercises; Health, Subjective; Quality of Life
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Masking Description: In the study, participants will be left unaware of whether they are in the study or control group (single-blind masking).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Study group intervention consists of a mobile application called "My Fight with Incontinence" structured according to the health belief model, and a 3-month follow-up.
  Interventions: Other: 3 months follow-up; Behavioral: Mobile application which named as "My Fighting with Incontinence"
- Control group (Other): In addition to routine care, control group intervention consists of the training booklet "My Fight with Incontinence" which includes healthy lifestyle behaviors, bladder training, and Kegel exercises related to urinary incontinence, and a 3-month follow-up.
  Interventions: Other: Training booklet prepared by the researchers on healthy lifestyle behaviors, bladder training, and Kegel exercises related to urinary incontinence.; Other: 3 months follow-up

INTERVENTIONS:
Other: Training booklet prepared by the researchers on healthy lifestyle behaviors, bladder training, and Kegel exercises related to urinary incontinence. — After the participants enrolled in the study, a training booklet prepared by the researchers on healthy lifestyle behaviors, bladder training, and Kegel exercises related to urinary incontinence will be given to the participants.
  Arms: Control group
Other: 3 months follow-up — Follow-ups will be made 3 times in total, on the basis of pre-test (baseline), intermediate follow-up test (6th week), and post-test (12th week).
Behavioral: Mobile application which named as "My Fighting with Incontinence" — The mobile application "My Fighting with Incontinence" aims to reduce incontinence symptoms of women with UI, ensure compliance with Kegel exercises, increase health belief and quality of life regarding UI and kegel exercises, and also allow researchers to be included in the awareness and management process.
  Arms: Study group

SUMMARY:
The first phase was designed in a methodological pattern in order to develop, usability, and performance of mobile application (mobileapp) called "My Fight with Incontinence". Aim of the second phase of the study was to evaluate the effect of mobileapp developed according to the health belief model on incontinence symptoms, Kegel exercise compliance, health belief and quality of life towards UI and kegel exercises in women with UI. The study was planned in a single-center, single-blind, one-to-one, parallel-group, randomized controlled trial design with a 3-month follow-up period. The research will be carried out in the Urology service and polyclinics of Eskişehir Osmangazi University Health Practice and Research Hospital. The study population of the research consists of 203 female patients over the age of 18 who were followed up with the diagnosis of Stress, Urge, and Mixed Type UI. Sample selection will not be made in the first stage of the study, and mobileapp will be tested on people aged 18 and over who can be reached, working, studying, or receiving treatment at Eskişehir Osmangazi University Training, Application and Research Hospital and Eskişehir Osmangazi University. The number of samples required for the study was determined by the power analysis made in the GPower 3.1 package program. Assuming that there may be losses during the follow-up and considering the possibility of nonparametric testing, a total of 96 individuals, 48 in each group, with an increase of 20%, will form the research group. In the second stage of the study, "Incontinence Severity Index Questionnaire", "International Urinary Incontinence Inquiry Form-Short Form (ICIQ-SF)", "Kegel Exercise Compliance Follow-up Form", "Health Belief Scale for Urinary Incontinence and Kegel Exercise", "Urogenital Distress Inventory-6 (UDI-6) and Incontinence Impact Questionnaire-7 (IIQ-7)" will be used. Control group will be given a training booklet called "My Fight with Incontinence", which includes healthy lifestyle behaviors, bladder training, and Kegel exercises related to UI after the pre-tests are applied. After pre-tests are applied to the study group, "My Fight with Incontinence" mobileapp will be installed on their mobile phones by researcher. Reminders will be sent to the patients on a regular basis via the mobileapp. Participants in both the control and study groups will be provided with the link of the survey form created via google forms in the 6th and 12th weeks by sending an SMS.

DETAILED DESCRIPTION:
Conservative, surgical, and pharmacological treatment methods are available in the treatment of urinary incontinence. Despite this, the first preferred method of treatment is the conservative treatment method. One of these methods and the most preferred one is pelvic floor muscle training (Kegel exercise). The reason why it is one of the most preferred treatment methods is that it is a reliable and effective method in reducing UI and increasing the quality of life. Research shows that mobile applications are effective in maintaining pelvic floor muscle exercise (Kegel exercise), improving quality of life, reducing urinary incontinence symptoms, accelerating the healing process, and facilitating access to care.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research
* Being a female
* Being in the age range of 18-65
* Using a smart mobile phone (for communicating via Whatsapp and installing a mobile application to the workgroup)
* BMI < 30kg/m2
* Being literate
* Having a diagnosis of urinary incontinence (stress, emergency/urge, mixed type)

Exclusion Criteria:

* Those who do not have an Android-based smartphone
* Have a physical or mental disability
* Those who have undergone vaginal and pelvic operations within 6 months
* Have given birth within 12 weeks
* Having a history of miscarriage within 6 weeks
* Those who have had recurrent vaginitis infections
* History of the cardiac implant or untreated cardiac arrhythmia
* Having a communication barrier

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only those who are biologically female will be included in the study.
Enrollment: 96 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline urinary incontinence severity at 6 weeks | 6th week
  The severity of the complaint of urinary incontinence will be evaluated using the "Incontinence Severity Index (ISI) Questionnaire". The lowest "1" and the highest "12" points can be obtained from the questionnaire. Accordingly, 1-2 points are evaluated as "mild", 3-6 points as "moderate", 8-9 points as "severe" and 12 points as "very severe".
Change from baseline urinary incontinence severity at 12 weeks | 12th week
  The severity of the complaint of urinary incontinence will be evaluated using the "Incontinence Severity Index (ISI) Questionnaire". The lowest "1" and the highest "12" points can be obtained from the questionnaire. Accordingly, 1-2 points are evaluated as "mild", 3-6 points as "moderate", 8-9 points as "severe" and 12 points as "very severe".
Change from the baseline level of urinary incontinence symptoms (frequency, amount, impact on daily life) at 6 weeks | 6th week
  "International urinary incontinence inquiry form-short form (ICIQ-SF)" will be used to evaluate urinary incontinence-related incontinence symptoms or complaints and their effect on the quality of life. The scale consists of 6 questions in total and 4 sub-dimensions as "frequency of urinary incontinence", "amount of urinary incontinence", "effect of urinary incontinence in daily life" and "causes of urinary incontinence". A minimum of 0 and a maximum of 21 points can be obtained from the scale. A high score on the scale indicates that urinary incontinence has a great impact on quality of life.
Change from the baseline level of urinary incontinence symptoms (frequency, amount, impact on daily life) at 12 weeks | 12th week
  "International urinary incontinence inquiry form-short form (ICIQ-SF)" will be used to evaluate urinary incontinence-related incontinence symptoms or complaints and their effect on the quality of life. The scale consists of 6 questions in total and 4 sub-dimensions as "frequency of urinary incontinence", "amount of urinary incontinence", "effect of urinary incontinence in daily life" and "causes of urinary incontinence". A minimum of 0 and a maximum of 21 points can be obtained from the scale. A high score on the scale indicates that urinary incontinence has a great impact on quality of life.
Change from baseline Kegel exercise compliance level at 6 weeks | 6th week
  The patients' compliance with kegel exercises (frequency of doing kegel exercises) will be evaluated with the "Kegel exercise compliance follow-up form" created by the researchers, in which the patients can mark the exercise practice times (7 days a week, morning-lunch-evening).
Change from baseline Kegel exercise compliance level at 12 weeks | 12th week
  The patients' compliance with kegel exercises (frequency of doing kegel exercises) will be evaluated with the "Kegel exercise compliance follow-up form" created by the researchers, in which the patients can mark the exercise practice times (7 days a week, morning-lunch-evening).
Change from baseline urinary incontinence quality of life at 6 weeks | 6th week
  Urogenital distress inventory-6 (UDI-6) and Incontinence effect questionnaire-7 (IIQ-7) will be used to determine the quality of life of patients with urinary incontinence. A minimum of 0 and a maximum of 18 points can be obtained from UDI-6, and a minimum of 0 and a maximum of 21 points can be obtained from IIQ-7. The total score of both forms is calculated at over 100 points. Low scores indicate higher quality of life.
Change from baseline urinary incontinence quality of life at 12 weeks | 12th week
  Urogenital distress inventory-6 (UDI-6) and Incontinence effect questionnaire-7 (IIQ-7) will be used to determine the quality of life of patients with urinary incontinence. A minimum of 0 and a maximum of 18 points can be obtained from UDI-6, and a minimum of 0 and a maximum of 21 points can be obtained from IIQ-7. The total score of both forms is calculated at over 100 points. Low scores indicate higher quality of life.
Change from baseline health belief level for urinary incontinence and kegel exercise at 6 weeks | 6th week
  "Health belief scale for urinary incontinence and kegel exercise" will be used to determine the beliefs of individuals about urinary incontinence and kegel exercise. The scale consists of 49 questions in 5-point Likert type and 6 sub-dimensions: "sensitivity", "seriousness", "health motivation", "kegel exercise benefit perception", "kegel exercise obstacle perception" and "self-efficacy". The scale does not have a total score. Sensitivity, seriousness, health motivation, kegel exercise benefit perception, and self-efficacy sub-dimensions are positive, while the kegel exercise obstacle perception sub-dimension is negative. Higher scores increase sensitivity, seriousness, and motivation; It means that benefits are perceived high for the perception of benefit, and obstacles are perceived high for the perception of obstacles.
Change from baseline health belief level for urinary incontinence and kegel exercise at 12 weeks | 12th week
  "Health belief scale for urinary incontinence and kegel exercise" will be used to determine the beliefs of individuals about urinary incontinence and kegel exercise. The scale consists of 49 questions in 5-point Likert type and 6 sub-dimensions: "sensitivity", "seriousness", "health motivation", "kegel exercise benefit perception", "kegel exercise obstacle perception" and "self-efficacy". The scale does not have a total score. Sensitivity, seriousness, health motivation, kegel exercise benefit perception, and self-efficacy sub-dimensions are positive, while the kegel exercise obstacle perception sub-dimension is negative. Higher scores increase sensitivity, seriousness, and motivation; It means that benefits are perceived high for the perception of benefit, and obstacles are perceived high for the perception of obstacles.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Duru, PhD, Principal Investigator — Department of Public Health Nursing, Eskisehir Osmangazi University, Turkey
Locations (1):
- Eskişehir Osmangazi University Health Practice and Research Hospital, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No